CLINICAL TRIAL: NCT06011824
Title: Megakaryocytes and Platelets, Harmful or Helpful in Breast Cancer Cell Metastasis
Brief Title: A Study of Effect of Megakaryocytes and Platelets in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-004958; NCI-2023-06775 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-08-08; First posted 2023-08-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Megakaryocytes; Platelets
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw. 10-12 mL total into lavender-top (EDTA) tubes, however up to 24 mL may be obtained should a redraw be needed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Biopsy Negative: Female age 18 and above with negative breast biopsy
  Interventions: Other: Blood draw
- Biopsy positive for carcinoma in situ (ductal, lobular, or other): Females age 18 and above with any subtype of breast cancer (ductal, lobular, or other)
  Interventions: Other: Blood draw
- Biopsy positive for Stage 1, 2, or 3 invasive carcinoma (ductal, lobular, or other): Females age 18 and above with any subtype of breast cancer (HER2+, ER/PR, TNBC, BRCA1 +/-, other).
  Interventions: Other: Blood draw
- Metastatic Stage IV: Females age 18 and above with any subtype of breast cancer, including metastases
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — 10-12mL of blood will be drawn one time, unless a redraw is needed, in which case up to 24 mL will be drawn (10-12 mL each draw)

SUMMARY:
Determining if Megakaryocytes and Platelets are Harmful or Helpful in Breast Cancer Cell Metastasis

DETAILED DESCRIPTION:
The purpose of this study is to determine how megakaryocytes (cells in the bone marrow responsible for making platelets, which are necessary for blood clotting) affect the survival and growth/division patterns of breast cancer stem cells, and the effects of breast cancer cells on megakaryocyte survival and function. Through chart review, the study team will look at the relationship between different blood components and different breast cancer diagnoses.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1-Biopsy negative

* Females age 18 and above

Cohort 2-Biopsy positive for carcinoma in situ (ductal, lobular, or other)

* Females age 18 and above
* Any subtype of breast cancer

Cohort 3-Biopsy positive for Stage 1, 2, or 3 invasive carcinoma (ductal, lobular, or other)

* Females age 18 and above
* Any subtype of breast cancer
* Have no distant metastases

Cohort 4-Stage 4 Metastatic Disease

* Females age 18 and above
* Any subtype of breast cancer

Exclusion Criteria:

* Previous diagnosis with a known platelet disorder such as: Bernard Soulier disease, Jacobsen syndrome, Lowe syndrome, Thrombocytopenia, Thrombotic thrombocytopenic pupura, Von Willebrand disease, or the equivalent. Any condition in which antiplatelet or anticoagulant therapy with one of the following medications is being prescribed: Clopidogrel (Plavix), Warfarin (Coumadin or Jantoven), Prasugrel (Effient), or Ticagrelor (Brilinta).

Cohort 1-Biopsy negative

* Males
* Females less than age 18

Cohort 2-Biopsy positive for carcinoma in situ (ductal, lobular, or other)

* Males
* Females less than age 18
* Currently undergoing neoadjuvant therapy

Cohort 3-Biopsy positive for Stage 1, 2, or 3 invasive carcinoma (ductal, lobular, or other)

* Males
* Females less than age 18
* Presence of distant metastases
* Currently undergoing neoadjuvant therapy

Cohort 4-Stage 4 Metastatic Disease

* Males
* Females less than age 18
* Currently undergoing neoadjuvant therapy
* Less than 30 days from last adjuvant treatment for Stage I-III Breast Cancer (may be on Trastuzumab, Pertuzumab, or endocrine therapy only for maintenance therapy from their prior breast cancer diagnosis)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females
Study Population: For the prospective study: 20 women after biopsy for suspicious mammogram findings, 10 women with newly diagnosed metastatic cancer.
  Subject population (children, adults, groups): Women undergoing biopsy or suspicious mammogram finds and newly diagnosed female metastatic breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Platelet Counts | Baseline
  Measure of the number of platelets in the blood, reported as platelets per microliter of blood.

SECONDARY OUTCOMES:
Mean Corpuscular Volume (MCV) | Baseline
  Measures the average size of red blood cells, reported as femtoliters (fl).
Lymphocyte to neutrophil ratio | Baseline
  Ratio between the neutrophil and lymphocyte counts measured in peripheral blood.
Levels of tumor educated platelets | Baseline
  Number of tumor educated platelets, measured by the analysis of cell surface markers for expression of certain markers such as VEGF, PDGFR, MMP1, TGFb, and or other cell adhesion molecules.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H. Okuno, M.D., Principal Investigator — Mayo Clinic Health System-Franciscan Healthcare
Locations (1):
- Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials